CLINICAL TRIAL: NCT01912729
Title: Technology Assisted Intervention for the Treatment and Prevention of Depression
Brief Title: Technology Assisted Programs That Promote Mental Health for Teenagers
Acronym: ProjectTECH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Mohr, Director, Center for Behavioral Intervention Technologies; Professor, Department of Preventive Medicine, Northwestern University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P20MH090318 STU00056069-FTPT; P20MH090318 (NIH)
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Results first posted 2018-11-21 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-11

CONDITIONS: Depression
Keywords: Depression prevention; Technology Assisted; Adolescents; Peer networked
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Networked Peer Support with Peer Guide (Experimental): Participants will have access to tools and lessons based on Cognitive Behavior Therapy through a mobile phone application. Additionally, participants will have access to a private social network that connects them with other participants in the study. The social network will be moderated by a trained peer coach.
  Interventions: Behavioral: Networked Peer Support with Peer Guide
- Networked Peer Support with Clinician Coach (Experimental): Participants will have access to tools and lessons based on Cognitive Behavior Therapy through a mobile phone application. Additionally, participants will have access to a private social network that connects them with other participants in the study. The social network will be moderated by a clinician coach.
  Interventions: Behavioral: Networked Peer Support with Clinician Coach
- Wait List Control (No Intervention): Participants may be asked to wait for up to 8 weeks until minimum group size is met. After 4 weeks from baseline, if a group has not yet started, we will conduct another assessment. These participants will serve as the Wait List Control group.

INTERVENTIONS:
Behavioral: Networked Peer Support with Peer Guide — Participants will have access to tools and lessons based on Cognitive Behavior Therapy through a web application that can be accessed on a smartphone or computer. Additionally, participants will have access to a private social network that connects them with other participants in the study. Participants will be supported by a peer guide. The peer guide will be another high school student around the same age as participants.
  Arms: Networked Peer Support with Peer Guide
Behavioral: Networked Peer Support with Clinician Coach — Participants will have access to tools and lessons based on Cognitive Behavior Therapy through a web application that can be accessed on a smartphone or computer. Additionally, participants will have access to a private social network that connects them with other participants in the study. Participants will be supported by a clinical psychologist.
  Arms: Networked Peer Support with Clinician Coach

SUMMARY:
The mission of this project is to develop novel systems of care that can provide efficacious, scalable, cost-effective, participant friendly behavioral intervention technologies (BITs) for the prevention of depression in adolescents. The investigators define BITs as interventions that use information and telecommunications technologies such as the internet, mobile or traditional phones, computers and/or other technologies to support and deliver psychological and behavioral interventions. Through usability testing, focus interviews, and field trials, investigators may modify the technologies and intervention based on immediate usage data.

DETAILED DESCRIPTION:
The mission of this project is to develop novel systems of care that can provide efficacious, scalable, cost-effective, participant friendly behavioral intervention technologies (BITs) for the prevention of depression in adolescents. The investigators define BITs as interventions that use information and telecommunications technologies such as the internet, mobile or traditional phones, computers and/or other technologies to support and deliver psychological and behavioral interventions. Through usability testing, focus interviews, and field trials, investigators may modify the technologies and intervention based on immediate usage data.

ELIGIBILITY:
Inclusion Criteria:

* Has a score of 12-39 (males) / 15-39 (females) on the Center for Epidemiologic Studies Depression Scale (CES-D) OR reported past month use of marijuana, cigarettes, alcohol or other substances on the Center for Disease Control Youth Risk Behavior Survey (YRBS).
* Is familiar with the use of computers and the Internet, as well as mobile phones
* Is able to speak and read English
* Is between 14-19 years of age

Exclusion Criteria:

* Is currently taking an antidepressant medication or has taken one in the previous 3 months
* Has visual, hearing, voice, or motor impairment that would prevent completion of study procedures or use of the Internet or mobile phone
* Is diagnosed with a psychotic disorder, bipolar disorder, dissociative disorder, current substance dependence, or other diagnosis for which participation in this trial is either inappropriate or dangerous. Inclusion of participants with symptoms of anxiety disorders, eating disorders and substance abuse disorders will be made on a case-by-case basis.
* Is severely suicidal (has ideation, plan, and intent in the past 12 months) .

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Mohr, Ph.D, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Networked Peer Support With Peer Guide | Networked Peer Support With Clinician Coach
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm 1 - Networked Peer Support With Peer Guide: Participants will have access to tools and lessons based on Cognitive Behavior Therapy through a mobile phone application. Additionally, participants will have access to a private social network that connects them with other participants in the study. The social network will be moderated by a trained peer coach.
  Networked Peer Support with Peer Guide: Participants will have access to tools and lessons based on Cognitive Behavior Therapy through a web application that can be accessed on a smartphone or computer. Additionally, participants will have access to a private social network that connects them with other participants in the study. Participants will be supported by a peer guide. The peer guide will be another high school student around the same age as participants.
- Arm 2 - Networked Peer Support With Clinician Coach: Participants will have access to tools and lessons based on Cognitive Behavior Therapy through a mobile phone application. Additionally, participants will have access to a private social network that connects them with other participants in the study. The social network will be moderated by a clinician coach.
  Networked Peer Support with Clinician Coach: Participants will have access to tools and lessons based on Cognitive Behavior Therapy through a web application that can be accessed on a smartphone or computer. Additionally, participants will have access to a private social network that connects them with other participants in the study. Participants will be supported by a clinical psychologist.
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Networked Peer Support With Peer Guide | Arm 2 - Networked Peer Support With Clinician Coach | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.45 (0.999) | 16.0 (0.94) | 16.23 (0.99)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 6 | 3 | 9
  Female | 13 | 16 | 29
  Other | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 16 | 13 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 12 | 12 | 24
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Program Logins Per Participant by Week.
Description: Program usage data were examined by number of logins per participant by week. Participants in the study tended to access the program multiple times and explored the program tools.
Time Frame: Weeks 1-8
Measure: Mean (Standard Deviation); unit: number of program logins
Arm/Group | Arm 1 - Networked Peer Support With Peer Guide | Arm 2 - Networked Peer Support With Clinician Coach
Number analyzed (Participants) | 20 | 19
number of program logins
  Week 1 | 9.15 (4.12) | 8.17 (4.02)
  Week 2 | 3.6 (2.91) | 6.06 (6.48)
  Week 3 | 2.8 (2.12) | 3.39 (2.62)
  Week 4 | 2.8 (2.44) | 2.44 (2.55)
  Week 5 | 2.6 (2.01) | 2.28 (1.87)
  Week 6 | 2.05 (1.9) | 2.33 (2.57)
  Week 7 | 1.7 (1.75) | 1.11 (1.84)
  Week 8 | 1.95 (2.31) | 1.22 (1.4)

2. Primary Outcome: USE (Usefulness, Satisfaction and Ease of Use) Questionnaire
Description: A modified version of the Usefulness, Satisfaction and Ease of use questionnaire (USE; Lund, 2001) was used, particularly regarding the participants' relationships with the peer network. The USE questionnaire is a 19 item measure of usability with 4 subscales: Usefulness, Ease of Learning, Ease of Use, and Satisfaction. The items are rated on 7 point Likert rating scales, with 1 = Strongly disagree to 7 = Strongly agree.
  Lund, A.M., 2001. Measuring Usability with the USE Questionnaire.
Time Frame: Week 4 and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 - Networked Peer Support With Peer Guide | Arm 2 - Networked Peer Support With Clinician Coach
Number analyzed (Participants) | 20 | 19
units on a scale
  Usefulness at Week 4 | 4.04 (1.73) | 4.4 (1.01)
  Usefulness at Week 8 | 4.36 (1.62) | 4.53 (0.97)
  Ease of Learning at Week 4 | 5.21 (2.07) | 5.55 (1.4)
  Ease of Learning at Week 8 | 5.73 (1.25) | 5.38 (1.53)
  Ease of Use at Week 4 | 4.79 (1.95) | 5.15 (1.28)
  Ease of Use at Week 8 | 4.96 (1.27) | 5.03 (1.44)
  Satisfaction at Week 4 | 4.18 (2.04) | 4.2 (1.44)
  Satisfaction at Week 8 | 4.23 (2.01) | 4.29 (1.27)

3. Primary Outcome: SUS (System Usability Scale) Questionnaire
Description: The SUS questionnaire is a 10 item measure that assesses usability, acceptability and satisfaction; each item has five response options for respondents, from 1 = Strongly disagree to 5 = Strongly agree. The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. Specifically, for odd items: subtract one from the user response. For even-numbered items: subtract the user responses from 5. This scales all values from 0 to 4 (with four being the most positive response). Add up the converted responses for each user and multiply that total by 2.5. This converts the range of possible values from 0 to 100 instead of from 0 to 40. A SUS score above a 68 would be considered above average and anything below 68 is below average.
Time Frame: Week 4 and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 - Networked Peer Support With Peer Guide | Arm 2 - Networked Peer Support With Clinician Coach
Number analyzed (Participants) | 20 | 19
units on a scale
  SUS score at Week 4 | 61.53 (15.1) | 71.91 (18.74)
  SUS score at Week 8 | 66.72 (14.82) | 69.53 (21.16)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Arm 1 - Networked Peer Support With Peer Guide | Arm 2 - Networked Peer Support With Clinician Coach
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes